CLINICAL TRIAL: NCT01217073
Title: A Phase IIb, Randomized, Placebo-Controlled, Dose-Range Finding Clinical Trial to Study the Safety and Efficacy of MK-3102 in Patients With Type 2 Diabetes Mellitus and Inadequate Glycemic Control
Brief Title: A Dose-Range Finding Study in Participants With Type 2 Diabetes (MK-3102-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-006; 2010-022193-13 (EudraCT Number); 2011-000656-42 (EudraCT Number)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Omarigliptin 0.25 mg (Base) (Experimental): Omarigliptin 0.25 mg administered once weekly for 12 weeks (Base)
  Interventions: Drug: Omarigliptin
- Omarigliptin 1 mg (Base) (Experimental): Omarigliptin 1 mg administered once weekly for 12 weeks (Base)
  Interventions: Drug: Omarigliptin
- Omarigliptin 3 mg (Base) (Experimental): Omarigliptin 3 mg administered once weekly for 12 weeks (Base)
  Interventions: Drug: Omarigliptin
- Omarigliptin 10 mg (Base) (Experimental): Omarigliptin 10 mg administered once weekly for 12 weeks (Base)
  Interventions: Drug: Omarigliptin
- Omarigliptin 25 mg (Base) (Experimental): Omarigliptin 25 mg administered once weekly for 12 weeks (Base)
  Interventions: Drug: Omarigliptin
- Placebo (Base) (Placebo Comparator): Matching placebo to omarigliptin administered once weekly for 12 weeks (Base)
  Interventions: Drug: Placebo to omarigliptin
- Pooled omarigliptin (Extension) (Experimental): Participants who received omarigliptin during the base study, received omarigliptin 25 mg once weekly and placebo to metformin once daily for 66 weeks (Extension).
  Interventions: Drug: Omarigliptin; Drug: Placebo to metformin
- Placebo/Metformin (Active Comparator): Participants who received matching placebo to omarigliptin during the base period, received pioglitazone administered once daily and matching placebo to omarigliptin once weekly for 66 weeks (extension period). Note: A protocol amendment removed pioglitazone during the extension period. Participants discontinued pioglitazone and switched to blinded metformin. Participants who were previously rescued with open-label metformin during the base period continued in the extension period on open-label metformin.
  Interventions: Drug: Placebo to omarigliptin; Drug: Pioglitazone; Drug: Metformin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin 0.25, 1, 1.5, 10 or 25 mg oral capsule administered once weekly. For omarigliptin 3 mg, participants received two omarigliptin 1.5 mg capsules.
  Arms: Omarigliptin 0.25 mg (Base); Omarigliptin 1 mg (Base); Omarigliptin 10 mg (Base); Omarigliptin 25 mg (Base); Omarigliptin 3 mg (Base); Pooled omarigliptin (Extension)
Drug: Placebo to omarigliptin — Matching placebo to omarigliptin 0.25, 1, 1.5, 10 or 25 mg oral capsule administered once weekly. For matching placebo to omarigliptin 3 mg, participants received two matching placebo to omarigliptin 1.5 mg capsules.
  Arms: Placebo (Base); Placebo/Metformin
Drug: Pioglitazone — Pioglitazone 15 mg oral tablet or capsule administered once daily
  Arms: Placebo/Metformin
Drug: Metformin — Metformin 500 mg oral tablet administered once or twice daily
  Arms: Placebo/Metformin
Drug: Placebo to metformin — Matching placebo to metformin oral tablet administered once daily
  Arms: Pooled omarigliptin (Extension)

SUMMARY:
The purpose of this study is to assess the hypothesis that treatment with study medication (omarigliptin; MK-3102) provides greater reduction in A1C Hemoglobin (a marker of diabetic severity) compared with placebo, after 12 weeks of treatment. The study will evaluate 5 different doses of omarigliptin to identify which dose is the most effective in the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
MK-3102-006-Ext 1 added a 66-week extension to the base study (MK-3102 P006) to assess the long-term safety and tolerability of omarigliptin. To be eligible for the extension, participants must complete the double-blind base study, must have had at least a 75% compliance with study drug during the base study and can not meet any of the criteria for discontinuation. Participants randomized to placebo in the base study will be switched in a blinded manner to pioglitazone 30 mg once daily, in the extension study prior to implementation of amendment P006-13. Once amendment P006-13 has been IRB/IEC approved and blinded metformin drug supply is available at the site, participants will be switched from pioglitazone to metformin, starting at 500 mg once daily and titrated up to 1000 mg twice daily. Participants with a contraindication to metformin will be discontinued from the study. Participants randomized to 0.25 mg, 1 mg, 3 mg, and 10 mg of omarigliptin in the base study will be switched to omarigliptin 25 mg; those randomized to 25 mg of omarigliptin in the base study will continue on the same dose in the extension study. After the clinical dose of omarigliptin selected for further development has been identified based upon the results of the base study, all participants randomized to omarigliptin will be switched to the identified clinical dose.

ELIGIBILITY:
Inclusion Criteria:

The prospective participant must meet, at least, all of the criteria below (among others determined by the study staff) to be eligible for study participation.

The participant:

* Has type 2 diabetes mellitus and is between 18 and 70 years of age; for Japan, 20 to 70 years of age;
* Has a body mass index (BMI) > 20 kg/m^2 and < 43 kg/m^2; for Japan: BMI >18 kg/m^2 and <43 kg/m^2;
* Is currently not on an antihyperglycemic agent (AHA) medication (off for ≥ 14 weeks) or is on oral AHA therapy but has inadequate glycemic control;
* Is a male, or a female who is highly unlikely to conceive.

Exclusion Criteria:

If the prospective participant meets any of the criteria below (among others determined by the study staff) they will NOT be eligible for study participation.

The participant:

* Has a history of type 1 diabetes mellitus or a history of ketoacidosis;
* Is on a weight loss program or has started a weight loss medication within the prior 8 weeks;
* Has required insulin therapy within 14 weeks prior to signing informed consent;
* Has a medical history of active liver disease (other than nonalcoholic hepatic steatosis), including chronic active hepatitis B or C, cirrhosis, or symptomatic gallbladder disease;
* Has congestive heart failure or has new or worsening signs or symptoms of coronary heart disease;
* Had any of the following disorders within the past 3 months: acute coronary syndrome, coronary artery intervention, stroke or transient ischemic neurological disorder;
* Has a history of malignancy or clinically important hematological disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2010-10-08 (Actual); Primary Completion 2012-01-03 (Actual); Study Completion 2013-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sheu WH, Gantz I, Chen M, Suryawanshi S, Mirza A, Goldstein BJ, Kaufman KD, Engel SS. Safety and Efficacy of Omarigliptin (MK-3102), a Novel Once-Weekly DPP-4 Inhibitor for the Treatment of Patients With Type 2 Diabetes. Diabetes Care. 2015 Nov;38(11):2106-14. doi: 10.2337/dc15-0109. Epub 2015 Aug 26. PMID 26310692
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3102-006&kw=3102-006&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Omarigliptin 0.25 mg (Base): Omarigliptin 0.25 mg administered once weekly for 12 weeks (base period)
- Omarigliptin 1 mg (Base): Omarigliptin 1 mg administered once weekly for 12 weeks (base period)
- Omarigliptin 3 mg (Base): Omarigliptin 3 mg administered once weekly for 12 weeks (base period)
- Omarigliptin 10 mg (Base): Omarigliptin 10 mg administered once weekly for 12 weeks (base period)
- Omarigliptin 25 mg (Base): Omarigliptin 25 mg administered once weekly for 12 weeks (base period)
- Placebo (Base): Matching placebo to omarigliptin administered once weekly for 12 weeks (base period)
- Pooled Omarigliptin (Extension): Participants received omarigliptin 25 mg once weekly and placebo to metformin once daily for 66 weeks (extension period)
- Placebo/Metformin (Extension): Participants who received matching placebo to omarigliptin during the base study, received pioglitazone 30 mg once daily and matching placebo to omarigliptin once weekly for 66 weeks (Extension period). Participants were switched from pioglitazone to metformin starting at 500 mg once daily and titrated up to 1000 mg twice a day
Period: Base Period
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base) | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Started | 113 | 115 | 114 | 115 | 114 | 114 | 0 | 0
Completed | 106 | 110 | 107 | 113 | 99 | 105 | 0 | 0
Not Completed | 7 | 5 | 7 | 2 | 15 | 9 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 0
Not completed — Alanine aminotransferase (ALT)/AST | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Excluded medication | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 5 | 1 | 5 | 5 | 0 | 0
Period: Extension Period
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base) | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 405 | 80
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 314 | 60
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 91 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 5
Not completed — ALT/AST | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Contraindication to study medication | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Creatinine/eGFR | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Excluded medication | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Site discontinued study participation | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 8

BASELINE CHARACTERISTICS:
Population: Population includes all participants randomized during the base period. The extension period only included participants who completed the base period and consented to enter the extension period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base) | Total
Number analyzed (Participants) | 113 | 115 | 114 | 115 | 114 | 114 | 685
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (8.9) | 55.7 (8.5) | 55.3 (8.5) | 54.4 (10.0) | 55.1 (8.5) | 55.9 (8.4) | 55.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 49 | 59 | 45 | 49 | 298
  Male | 65 | 67 | 65 | 56 | 69 | 65 | 387
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] — Participants with data: Omariglptin 0.25 mg, n=113; Omariglptin 1 mg, n=115; Omariglptin 3 mg, n=114; Omariglptin 10 mg, n=115; Omariglptin 25 mg, n=113; Placebo, n=113; Total, n=683
  Percent | 8.1 (0.9) | 8.0 (0.9) | 7.9 (0.9) | 8.0 (0.9) | 8.1 (1.0) | 8.1 (0.9) | 8.1 (0.9)
2-hour post meal glucose (2-hr PMG) [Mean (Standard Deviation); unit: mg/dL] — Participants with data: Omariglptin 0.25 mg, n=111; Omariglptin 1 mg, n=113; Omariglptin 3 mg, n=113; Omariglptin 10 mg, n=112; Omariglptin 25 mg, n=111; Placebo, n=110; Total, n=670
  mg/dL | 229.4 (63.7) | 229.3 (64.5) | 234.7 (81.7) | 231.6 (72.3) | 245.3 (82.7) | 241.4 (72.2) | 235.2 (73.2)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Participants with data: Omariglptin 0.25 mg, n=113; Omariglptin 1 mg, n=115; Omariglptin 3 mg, n=114; Omariglptin 10 mg, n=115; Omariglptin 25 mg, n=114; Placebo, n=113; Total, n=684
  mg/dL | 170.3 (45.3) | 169.4 (42.4) | 169.0 (42.6) | 166.8 (37.6) | 173.9 (47.6) | 171.9 (42.8) | 170.2 (43.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma A1C Levels at Week 12
Description: A1C levels were measured as a percent. Change from baseline was calculated by subtracting the baseline level from the Week 12 level.
Time Frame: Baseline (Week 0) and Week 12
Population: Full analysis set defined as all randomized participants who received at least one dose of study treatment and had a baseline measurement or a post-randomization measurement for the analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base)
Number analyzed (Participants) | 113 | 115 | 114 | 115 | 114 | 113
Percent | -0.14 [-0.30 to 0.01] | -0.36 [-0.51 to -0.20] | -0.35 [-0.50 to -0.19] | -0.53 [-0.68 to -0.38] | -0.57 [-0.73 to -0.42] | 0.14 [-0.01 to 0.29]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — With terms for treatment, prior AHA therapy status, geographic region (Japan/ex-Japan), and the interaction of time by treatment, time by prior AHA therapy status, with the constraint that the mean baseline is the same for all treatment groups; Difference in least squares mean = -0.71, 95% CI 2-sided [-0.93 to -0.50]
Statistical Analysis 2: Comparison: Omarigliptin 10 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -0.67, 95% CI 2-sided [-0.88 to -0.45]
Statistical Analysis 3: Comparison: Omarigliptin 3 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -0.49, 95% CI 2-sided [-0.70 to -0.27]
Statistical Analysis 4: Comparison: Omarigliptin 1 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -0.50, 95% CI 2-sided [-0.71 to -0.28]
Statistical Analysis 5: Comparison: Omarigliptin 0.25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p = 0.012, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -0.28, 95% CI 2-sided [-0.50 to -0.06]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event During the Base Period
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the Sponsor's product, is also an adverse event. Data presented below excludes data after the initiation of glycemic rescue.
Time Frame: Up to 16 weeks (including 28 days following the last dose of study drug)
Population: The all participants as treated population defined as all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received during the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base)
Number analyzed (Participants) | 113 | 115 | 114 | 115 | 114 | 113
Percentage of participants | 37.2 | 43.5 | 36.8 | 36.5 | 33.3 | 31.0
Statistical Analysis 1: Comparison: Omarigliptin 0.25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 6.2, 95% CI 2-sided [-6.2 to 18.4]
Statistical Analysis 2: Comparison: Omarigliptin 1 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 12.5, 95% CI 2-sided [-0.1 to 24.7]
Statistical Analysis 3: Comparison: Omarigliptin 3 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 5.9, 95% CI 2-sided [-6.5 to 18.0]
Statistical Analysis 4: Comparison: Omarigliptin 10 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 5.5, 95% CI 2-sided [-6.8 to 17.7]
Statistical Analysis 5: Comparison: Omarigliptin 25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 2.4, 95% CI 2-sided [-9.8 to 14.5]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event During the 12-week Base Period
Description: as for outcome 2
Time Frame: Up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base)
Number analyzed (Participants) | 113 | 115 | 114 | 115 | 114 | 113
Percentage of participants | 0.9 | 0 | 0.9 | 0 | 3.5 | 0.9
Statistical Analysis 1: Comparison: Omarigliptin 0.25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 0.0, 95% CI 2-sided [-4.1 to 4.1]
Statistical Analysis 2: Comparison: Omarigliptin 1 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = -0.9, 95% CI 2-sided [-4.9 to 2.4]
Statistical Analysis 3: Comparison: Omarigliptin 3 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 0.0, 95% CI 2-sided [-4.1 to 4.0]
Statistical Analysis 4: Comparison: Omarigliptin 10 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = -0.9, 95% CI 2-sided [-4.9 to 2.4]
Statistical Analysis 5: Comparison: Omarigliptin 25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; Difference in percentage = 2.6, 95% CI 2-sided [-1.7 to 7.9]

4. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event During the 66-week Extension Period
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the Sponsor's product, is also an adverse event. Data presented below excludes data after the initiation of glycemic rescue.
Time Frame: Up to 70 Weeks (Weeks 12 to 78 plus 4-week follow-up period)
Population: Analysis population defined as all randomized participamts who received at least one dose of extension study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received. Participants who received glycemic rescue during the base period were excluded from this analysis population.
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Omarigliptin (Extension): Participants received omarigliptin 25 mg once weekly for 66 weeks (extension period)
Arm/Group | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Number analyzed (Participants) | 392 | 76
Percentage of participants | 66.8 | 65.8
Statistical Analysis 1: Comparison: Pooled Omarigliptin (Extension) vs Placebo/Metformin (Extension); Test type: Superiority or Other; Difference in percent = 1.0, 95% CI 2-sided [-9.8 to 13.1]

5. Primary Outcome: Percentage of Participants Who Discontinued From Study Drug Due to an Adverse Event During the 66-week Extension Period
Description: as for outcome 4
Time Frame: Up to 66 weeks (Weeks 12 to 78)
Population: Analysis population defined as all randomized participants who received at least one dose of extension study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received. Participants who received glycemic rescue during the base period were excluded from this analysis population.
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Number analyzed (Participants) | 392 | 76
Percentage of participants | 3.8 | 5.3
Statistical Analysis 1: Comparison: Pooled Omarigliptin (Extension) vs Placebo/Metformin (Extension); Test type: Superiority or Other; Difference in percent = -1.4, 95% CI 2-sided [-9.1 to 2.6]

6. Secondary Outcome: Change From Baseline in 2 Hour-post-meal Glucose (2h-PMG) Levels at Week 12
Description: Change from baseline was calculated by subtracting the baseline level from the Week 12 level.
Time Frame: Baseline (Week 0) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base)
Number analyzed (Participants) | 112 | 113 | 114 | 114 | 112 | 111
mg/dL | -11.3 [-21.5 to -1.1] | -26.0 [-35.8 to -16.2] | -27.5 [-37.3 to -17.8] | -34.0 [-43.7 to -24.3] | -37.3 [-47.6 to -27.1] | 7.5 [-2.6 to 17.7]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -44.9, 95% CI 2-sided [-59.0 to -30.7]
Statistical Analysis 2: Comparison: Omarigliptin 10 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -41.6, 95% CI 2-sided [-55.3 to -27.8]
Statistical Analysis 3: Comparison: Omarigliptin 3 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -35.1, 95% CI 2-sided [-48.9 to -21.3]
Statistical Analysis 4: Comparison: Omarigliptin 1 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -33.5, 95% CI [-47.3 to -19.7]
Statistical Analysis 5: Comparison: Omarigliptin 0.25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p = 0.009, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -18.8, 95% CI 2-sided [-32.9 to -4.8]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Levels at Week 12
Description: Change from baseline was calculated by subtracting the baseline level from the Week 12 level.
Time Frame: Baseline (Week 0) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base)
Number analyzed (Participants) | 113 | 115 | 114 | 115 | 114 | 113
mg/dL | 1.2 [-4.5 to 7.0] | -15.3 [-20.9 to -9.7] | -10.6 [-16.3 to -4.8] | -9.8 [-15.4 to -4.2] | -17.7 [-23.5 to -11.8] | 3.7 [-2.0 to 9.4]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -21.4, 95% CI 2-sided [-29.4 to -13.4]
Statistical Analysis 2: Comparison: Omarigliptin 10 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -13.5, 95% CI 2-sided [-21.3 to -5.7]
Statistical Analysis 3: Comparison: Omarigliptin 3 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -14.3, 95% CI 2-sided [-22.2 to -6.3]
Statistical Analysis 4: Comparison: Omarigliptin 1 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -19.0, 95% CI 2-sided [-26.9 to -11.2]
Statistical Analysis 5: Comparison: Omarigliptin 0.25 mg (Base) vs Placebo (Base); Test type: Superiority or Other; p = 0.539, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 1]; Difference in least squares mean = -2.5, 95% CI 2-sided [-10.4 to 5.5]

8. Secondary Outcome: Mean Plasma A1C Level at Baseline of the Extension Period
Description: A1C levels were measured as a percent at baseline (Week 0) for participants who entered the extension period.
Time Frame: Baseline (Week 0)
Population: All participants who entered the extension period of the study with available A1C baseline data.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Number analyzed (Participants) | 404 | 80
Percent | 8.0 (0.9) | 8.2 (0.9)

9. Secondary Outcome: Change From Baseline in Plasma A1C Levels at Week 78
Description: A1C levels were measured as a percent. Change from baseline was calculated by subtracting the baseline level from the Week 78 level.
Time Frame: Baseline (Week 0) and Week 78
Population: Extension full analysis set population defined as all randomized participants who received at least one dose of extension study treatment, have baseline and at least one post-randomization observation for the analysis endpoint subsequent to at least one dose of extension study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Omarigliptin 0.25 mg (Base)/25 mg (Extension): Omarigliptin 0.25 mg administered once weekly for 12 weeks (Base) followed by omarigliptin 25 mg once weekly for 66 weeks (Extension)
- Omarigliptin 1 mg (Base)/25 mg (Extension): Omarigliptin 1 mg administered once weekly for 12 weeks (Base) followed by omarigliptin 25 mg once weekly for 66 weeks (Extension)
- Omarigliptin 3 mg (Base)/25 mg (Extension): Omarigliptin 3 mg administered once weekly for 12 weeks (Base) followed by omarigliptin 25 mg once weekly for 66 weeks (Extension)
- Omarigliptin 10 mg (Base)/25 mg (Extension): Omarigliptin 10 mg administered once weekly for 12 weeks (Base) followed by omarigliptin 25 mg once weekly for 66 weeks (Extension)
- Omarigliptin 25 mg (Base)/25 mg (Extension): Omarigliptin 25 mg administered once weekly for 12 weeks (Base) followed by omarigliptin 25 mg once weekly for 66 weeks (Extension)
- Placebo (Base)/Metformin (Extension): Matching placebo to omarigliptin administered once weekly for 12 weeks (Base) followed by pioglitazone 30 mg administered once daily and matching placebo to omarigliptin once weekly for 66 weeks (Extension). Piogliatazone was removed by a protocol amendment and replaced with metformin starting dose 500 mg one daily up-titrated to 1000 mg twice daily.
Arm/Group | Omarigliptin 0.25 mg (Base)/25 mg (Extension) | Omarigliptin 1 mg (Base)/25 mg (Extension) | Omarigliptin 3 mg (Base)/25 mg (Extension) | Omarigliptin 10 mg (Base)/25 mg (Extension) | Omarigliptin 25 mg (Base)/25 mg (Extension) | Placebo (Base)/Metformin (Extension)
Number analyzed (Participants) | 83 | 91 | 79 | 82 | 70 | 80
Percent | -0.57 [-0.89 to -0.25] | -0.55 [-0.85 to -0.26] | -0.30 [-0.62 to 0.02] | -0.60 [-0.93 to -0.28] | -0.46 [-0.80 to -0.11] | -0.88 [-1.19 to -0.57]

10. Secondary Outcome: Mean 2h-PMG Level at Baseline of the Extension Period
Description: Plasma 2h-PMG levels were measured at baseline (Week 0) for participants who entered the extension period.
Time Frame: Baseline (Week 0)
Population: All participants who entered the extension period of the study with available 2h-PMG baseline data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Number analyzed (Participants) | 402 | 79
mg/dL | 232.8 (69.5) | 244.5 (70.1)

11. Secondary Outcome: Change From Baseline in 2h-PMG at Week 78
Description: Change from baseline was calculated by subtracting the baseline level from the Week 78 level.
Time Frame: Baseline (Week 0) and Week 78
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 0.25 mg (Base)/25 mg (Extension) | Omarigliptin 1 mg (Base)/25 mg (Extension) | Omarigliptin 3 mg (Base)/25 mg (Extension) | Omarigliptin 10 mg (Base)/25 mg (Extension) | Omarigliptin 25 mg (Base)/25 mg (Extension) | Placebo (Base)/Metformin (Extension)
Number analyzed (Participants) | 83 | 91 | 79 | 82 | 70 | 79
mg/dL | -37.0 [-54.1 to -20.0] | -21.3 [-38.2 to -4.4] | -18.0 [-35.9 to -0.1] | -27.6 [-46.3 to -8.9] | -43.2 [-62.0 to -24.4] | -40.3 [-58.1 to -22.6]

12. Secondary Outcome: Mean FPG Level at Baseline of the Extension Period
Description: Plasma FPG levels were measured at baseline (Week 0) for particiapnts who entered the extension period.
Time Frame: Baseline (Week 0)
Population: All participants who entered the extension period of the study with available FPG baseline data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Number analyzed (Participants) | 405 | 80
mg/dL | 169.4 (41.7) | 172.9 (43.5)

13. Secondary Outcome: Change From Baseline in FPG Levels at Week 78
Description: Change from baseline was calculated by subtracting the baseline level from the Week 78 level.
Time Frame: Baseline (Week 0) and Week 78
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 0.25 mg (Base)/25 mg (Extension) | Omarigliptin 1 mg (Base)/25 mg (Extension) | Omarigliptin 3 mg (Base)/25 mg (Extension) | Omarigliptin 10 mg (Base)/25 mg (Extension) | Omarigliptin 25 mg (Base)/25 mg (Extension) | Placebo (Base)/Metformin (Extension)
Number analyzed (Participants) | 83 | 91 | 79 | 82 | 70 | 80
mg/dL | -7.4 [-22.4 to 7.6] | -11.3 [-25.0 to 2.5] | -2.0 [-17.1 to 13.1] | -10.0 [-25.0 to 5.0] | -0.7 [-16.7 to 15.3] | -19.6 [-34.1 to -5.1]

ADVERSE EVENTS:
Time Frame: Up to 82 weeks (including 28 days following the last dose of study drug)
Description: All participants as treated population. Serious AEs and non-serious AEs (NSAEs) include and exclude data after glycemic rescue, respectively. During the base period, 17 participants initiated glycemic rescue and were not included in the total number at risk for NSAEs during the extension period. MedDRA 15.1 was used for extension arms only.
Arm/Group | Omarigliptin 0.25 mg (Base) | Omarigliptin 1 mg (Base) | Omarigliptin 3 mg (Base) | Omarigliptin 10 mg (Base) | Omarigliptin 25 mg (Base) | Placebo (Base) | Pooled Omarigliptin (Extension) | Placebo/Metformin (Extension)
Serious Adverse Events (participants affected / at risk) | 0/113 | 1/115 | 0/114 | 2/115 | 3/114 | 0/113 | 28/405 | 3/80
Other Adverse Events (participants affected / at risk) | 6/113 | 7/115 | 4/114 | 5/115 | 7/114 | 6/113 | 76/392 | 10/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 0.25 mg (Base) (N=113) | Omarigliptin 1 mg (Base) (N=115) | Omarigliptin 3 mg (Base) (N=114) | Omarigliptin 10 mg (Base) (N=115) | Omarigliptin 25 mg (Base) (N=114) | Placebo (Base) (N=113) | Pooled Omarigliptin (Extension) (N=405) | Placebo/Metformin (Extension) (N=80)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 0.25 mg (Base) (N=113) | Omarigliptin 1 mg (Base) (N=115) | Omarigliptin 3 mg (Base) (N=114) | Omarigliptin 10 mg (Base) (N=115) | Omarigliptin 25 mg (Base) (N=114) | Placebo (Base) (N=113) | Pooled Omarigliptin (Extension) (N=392) | Placebo/Metformin (Extension) (N=76)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 13 (18) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (5) | 4 (4) | 4 (4) | 6 (6) | 4 (4) | 45 (52) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 23 (49) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.